CLINICAL TRIAL: NCT04840277
Title: Remote Hearing Aid Adjustment for Experienced Hearing Aid Users; a Randomised Controlled Trial
Brief Title: Remote Hearing Aid Adjustment for Experienced Hearing Aid Users
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sodra Alvsborgs Hospital (Other)
Responsible Party: Principal Investigator, Milijana Malmberg, PhD, audiologist, Sodra Alvsborgs Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Remote HA-fitting
Record Dates: First submitted 2021-03-29; First posted 2021-04-09 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Hearing Aids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Remote hearing aid adjustment. All participants in this group are offered hearing aids possible to adjust remotely.
  Interventions: Device: Remote hearing aid adjustment
- Control group (No Intervention): Traditional hearing aid adjustment

INTERVENTIONS:
Device: Remote hearing aid adjustment — The intervention group is offered remote hearing aid adjustment whilst the control group is offered traditional hearing aid adjustment the requires physical appointments at the clinic. Remote hearing aid adjustment is applicable through mobile applications that hearing aid users download to their mobile phones.
  Arms: Intervention group

SUMMARY:
Many hearing aid users experience substantial communication difficulties that may affect their participation in daily life situations negatively. One of the reasons for experiencing remaining problems could be due to unrealistic expectations, another reason could be that the hearing aid is not well adjusted or that the hearing aid user didn't got sufficient support and follow-up from the audiologist.

The purpose of this project is to offer remote hearing aid adjustment as an additional support for experienced hearing aid users.

ELIGIBILITY:
Inclusion Criteria:

* >18 yr of age
* experienced hearing aid user

Exclusion Criteria:

* <18 yr of age
* new hearing aid users

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Hearing Handicap Inventory for the Elderly/Adults (HHIE/A) | Change" is being assessed: at baseline, directly after completed rehabilitation, 6 months post and 1 year post
  Assessing emotional and social outcomes of a hearing loss; minimum 0 points to maximum 100 points, a higher score means worse outcome.

SECONDARY OUTCOMES:
The Abbreviated Profile of Hearing Aid Benefit (APHAB) | Change" is being assessed: at baseline, directly after completed rehabilitation, 6 months post and 1 year post
  Measures subjective hearing loss in four typical hearing situations; minimum

CONTACTS AND LOCATIONS:
Overall Officials: Milijana Malmberg, PhD, Principal Investigator — Hearing Organization, Sweden
Locations (1):
- Hearing Clinic, Hearing Organization, Borås, Vastra Gotalandsregion, Sweden

IPD SHARING:
Plan to Share IPD: No